CLINICAL TRIAL: NCT04415294
Title: Evaluating a Novel, Self-administered Device ("Flicker-App") That Measures Critical Flicker Frequency as a Test for Minimal Hepatic Encephalopathy in Cirrhosis
Brief Title: Flicker App for Minimal Hepatic Encephalopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, George Ioannou, Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00004521; R21DK117431 (NIH)
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Critical flicker frequency — Measure the critical flicker frequency as a screening test for hepatic encephalopathy using a portable self administered device

SUMMARY:
There is a great unmet clinical need for improved screening for MHE in patients with cirrhosis. We will demonstrate that the Flicker-App can be used in clinic as well as at home by patients with cirrhosis to measure CFF, a proven screening test for MHE. We will optimize the protocol, software, and hardware of the Flicker-App to create a product appropriate for production and distribution to patients

DETAILED DESCRIPTION:
SA 1. Determine whether cirrhotic patients (n=75) can self-administer the Flicker-App in clinic supervised by a research assistant and calculate the level of agreement between the CFF determined by the Flicker-App, the CFF determined by the "gold-standard" FFS device, and the test scores on the EncephalApp Stroop test.

SA 2. Determine whether cirrhotic patients (n=75) can self-administer the Flicker-App at home, including daily measurements over 1 week and weekly measurements over 6 weeks, and calculate the adherence to this protocol and the variability of these CFF measurements.

SA3. Make any necessary software or hardware adjustments to the Flicker-App to facilitate and simplify its self-administration by patients based on structured interview-questionnaires with the study participants and with clinical Gastroenterologists/Hepatologists

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis (standard criteria)
* Chronic liver disease

Exclusion Criteria:

* Grade III or IV hepatic encephalopathy
* Mini-mental state examination score ≤25 (suggestive of dementia)
* alcohol or illicit drug use within 3 months
* current use of benzodiazepines
* antiepileptics or psychotropic drugs
* color blindness
* severe vision impairment (blindness, macular degeneration).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhosis patients without Grade III or IV OHE
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
CFF Agreement | 1 day
  Level of agreement between Flicker App CFF and gold-standard device

CONTACTS AND LOCATIONS:
Overall Officials: George N Ioannou, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States